CLINICAL TRIAL: NCT05502055
Title: Perspectives on Healthcare Access and Equity of People With Parkinson's Disease Identifying as Lesbian, Gay, Bisexual, Transgender, Questioning, Intersex, or Two-spirit
Brief Title: Perspectives on Healthcare Access and Equity of People With Parkinson's Disease Identifying as LGBTQ+
Acronym: LGBTQ+_PD
Status: Suspended | Type: Observational
Why Stopped: Medical event of PI
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Tara McIsaac, Professor, Creighton University
Other Study IDs: 2003114-01
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Sexual Orientation
MeSH Terms: conditions — Parkinson Disease; Sexual Behavior | interventions — Focus Groups; Health Care Surveys

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- LGBTQ+_PD: Individuals who identify as LGBTQ+ and are diagnosed with PD
  Interventions: Other: Individual interviews; Other: Focus Groups; Other: National Survey
- Non-LGBTQ_PD: Individuals who identify as non-LGBTQ+ and are diagnosed with PD
  Interventions: Other: Individual interviews; Other: Focus Groups; Other: National Survey
- Care Partner: Individuals who are Care Partners of individuals with PD
  Interventions: Other: Individual interviews; Other: Focus Groups; Other: National Survey
- Health Care Provider: Health Care Providers who provide service to people with PD
  Interventions: Other: Individual interviews; Other: Focus Groups; Other: National Survey

INTERVENTIONS:
Other: Individual interviews — One on One interviews by Zoom video conferencing, < 2 hours in duration
Other: Focus Groups — Focus Groups discussions by Zoom video conferencing, < 2 hours in duration
Other: National Survey — Survey conducted online and distributed nationally

SUMMARY:
Study Rationale:

Older adults who identify as lesbian, gay, bisexual, transgender, or queer (LGBTQ+) have worse health than non-LGBTQ+ older adults. They and their care partners face greater barriers to getting healthcare and support from friends and family. This is because of lifelong stigma, discrimination, and isolation often separated from their families. Parkinson disease (PD) is a disease that usually appears in older age, so there may be many LGBTQ+ elders with PD, but there is currently no information on how people with PD who are LGBTQ+ are coping with their disease and aging. This study will begin to clarify their needs.

Hypothesis/Research Question:

What are the experiences and perspectives of LGBTQ+ people living with PD, their care partners, and physicians managing people with PD?

Study Design:

The investigators will interview 20 people with PD, half who identify as LGBTQ+ and half who are not. The investigators will also interview their care partners and physicians who treat people with PD. From the responses to the interview questions, investigators will create a survey that will be sent to people across the country.

Impact on Diagnosis/Treatment of Parkinson's Disease:

By understanding what LGBTQ+ people with PD need, and what ideas they have for improving their healthcare, better systems for meeting their needs can be built.

Next Steps for Development:

With this understanding, future work can focus on educating healthcare providers and clinics to improve the ways they talk with and treat LGBTQ+ people with PD.

DETAILED DESCRIPTION:
This mixed-methods study has a qualitative study component (1) and a quantitative study component (2):

Component 1) using a phenomenological inductive approach and Grounded Theory methodology the investigators will find and build themes from semi-structured interviews and focus groups with a) LGBTQ+ and non-LGBTQ+ individuals with PD, b) their care partners, and c) physicians to identify the experiences and perspectives on their health care and participation in research.

Component 2) survey development informed by results of Component 1, national distribution, and analysis of LGBTQ+ and non-LGBTQ+ people with PD, their caregivers and physicians, on barriers and access to health and disease information, healthcare delivery and participation in research.

The investigators plan to recruit 10 LGBTQ+ individuals with PD, 10 Non-LGBTQ+ individuals with PD, 10 care partners, and 10 healthcare providers for individual interviews, and 50 LGBTQ+ older adults with PD and care partners for focus groups consisting of 6-8 individuals each. For the national electronic survey investigators estimate needing a the sample size of approximately 380 responses calculated using a 95% confidence level (Z score=1.96), a standard deviation of .5, a 5% margin of error, and a population of 30,000. Purposive and Snowball sampling methods (nonprobability sampling) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PD
* Care partner of someone diagnosed with PD
* Health Care Provider providing services to individuals with PD
* Identify as LGBTQ+
* Identify as Non-LGBTQ+

Exclusion Criteria:

* Non-English speaking
* Inability to communicate via video conferencing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals from across the United States, from urban and rural areas and across diverse socioeconomic environments, with online access for a 2-hour period on a single day.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Themes of Lived Experience Accessing Health Care Services | 2 hours
  Inductive and iterative thematic analysis of transcripts
Themes of Lived Experience Providing Health Care Services to LGBTQ+ people with PD | 2 hours
  Inductive and iterative thematic analysis of transcripts

CONTACTS AND LOCATIONS:
Overall Officials: Tara L McIsaac, PT, PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No